CLINICAL TRIAL: NCT03968185
Title: Interfascial Infiltration to Relieve Functional Impairment in Patients Presenting to the Emergency Department for Acute Unspecific Low Back Pain: a Prospective Comparative Feasibility Study
Brief Title: Interfascial Infiltration for Acute Unspecific Low Back Pain in the Emergency Department
Acronym: PreSosLumbago
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0129
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Low Back Pain; Acute
Keywords: Low back pain; Pain; Disability; Interfascial infiltration; Anti-Inflammatory Agents, Non-Steroidal; Analgesics; Emergency department / emergency room / emergency management
MeSH Terms: conditions — Low Back Pain; Pain; Emergencies | interventions — Analgesics; Analgesics, Opioid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interfascial infiltration: Injection of L-bupivacaine (50 mg) and dexamethasone (4 mg) in the interfascial space under ultrasound guidance.
  Interventions: Other: Interfascial infiltration
- Standard medical treatment: Standard medical treatment include acetaminophen, NSAIDs and muscle relaxant as first line pharmacological treatment and escalation to analgesics level II or morphine if required, as needed for low back pain, in agreement with national guidelines Route of administration (orally or iv) was let at the discretion of the attending emergency physician.
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Other: Interfascial infiltration — Injection of L-bupivacaine (50 mg) and dexamethasone (4 mg) in the interfascial space under ultrasound guidance.
  Patients were kept under surveillance for at least one hour before discharge.
  Patients were discharged home with a 7 day supply of acetaminophen 1000 mg orally every 6 h, ketoprofen 100 mg, orally twice a day, and muscle relaxant as needed. Patients were instructed to take tramadol 50 mg, orally every 6h as needed for low back pain, in case of insufficient relief.
  Other Names: Interfascial injection
  Groups: Interfascial infiltration
Other: Standard medical treatment — Standard medical treatment include acetaminophen, NSAIDs and muscle relaxant as first line pharmacological treatment and escalation to analgesics level II or morphine if required, as needed for low back pain, in agreement with national guidelines Route of administration (orally or iv) was let at the discretion of the attending emergency physician.
  Patients were kept under surveillance for one hour before discharge. Patients were discharged home with a 7 day supply of acetaminophen 1000 mg orally every 6h, ketoprofen 100 mg, orally twice a day, and muscle relaxant as needed. Patients were instructed to take tramadol 50 mg, orally every 6h as needed for low back pain, in case of insufficient relief.
  Other Names: Analgesic, level I and II, opioid
  Groups: Standard medical treatment

SUMMARY:
Pain relief and functional impairment have been shown to remain poor to moderate over weeks after emergency department discharge, in patients who seek ED management for acute nontraumatic, nonradicular low back pain.

The investigators made the hypothesis that ultrasound-guided interfascial infiltration of local anesthesics and corticoid is efficient and safe in treating patients presenting to the ED with acute non specific low back pain. The investigators aimed to compare early and short term functional impairment and pain relief one day and 1 week after interfacial infiltration, as compared to standard medical treatment

DETAILED DESCRIPTION:
This is a single center observational feasibility study enrolling ED patients presenting with acute unspecific low back pain.

Ultrasound-guided interfascial infiltration is proposed to eligible patients presenting to our ED with low back pain and disability, as part of routine care. Patients receive standard medical treatment if they refuse interfascial infiltration or in case of absence or unavailability of a trained operator.

Patients were followed-up at 1 day and 7-days pots ED discharge by telephone interview conducted by an independent member of our research team not involved in patient's management

ELIGIBILITY:
Inclusion Criteria:

* adults aged between 18 and 70 years old
* presenting to the ED for low back pain from musculoskeletal origin, with symptoms evolving for less than 6 weeks,
* a score of 3 or more in the numeric pain scale (0-10)
* a score of 5 or greater on the Rolland Morris Disability Questionary (scale 0-24, RMDQ).

Exclusion Criteria:

* Traumatic or radicular pain or low back pain from alternative etiology
* allergy to local anesthetics
* Blood coagulation disorders
* Patients for whom follow-up by telephone interview was not possible
* Patients already enrolled in the study

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult emergency room patient as part of the usual management for non-traumatic, non-radicular, non-radicular, musculoskeletal pain with functional impotence defined by a score of 5 or higher on the EIFEL scale
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Improvement in functional impairment | 1 day
  Improvement in functional impairment as measured on the Roland-Morris Disability Questionnaire (RMQD), ranging from 0 no functional impairment to 24 severe disability

OTHER OUTCOMES:
Improvement in functional impairment | 7 days
  Improvement in functional impairment as measured on the Roland-Morris Disability Questionnaire (RMQD), ranging from 0 no functional impairment to 24 severe disability
improvement in pain score | 1 hour
  improvement in pain score as measured on a numeric pain scale (10 point- scale ranging from 0-no pain to 10-greatest pain)
improvement in pain score | 1 day
  improvement in pain score as measured on a numeric pain scale (10 point- scale ranging from 0-no pain to 10-greatest pain)
improvement in pain score as | 7 days
  improvement in pain score as measured on a numeric pain scale (10 point- scale ranging from 0-no pain to 10-greatest pain)
Pain Medicine consumption | 7 days
  Pain Medicine consumption within a week from ED management.
subsequent physician or other health professional visit related to low back pain | 7 days
  subsequent physician or other health professional visit related to low back pain within a week from ED management.

CONTACTS AND LOCATIONS:
Overall Officials: Mustapha Sebbane, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC